CLINICAL TRIAL: NCT02231515
Title: A Prospective, Randomized, Controlled Study to Assess Efficacy,Safety, and Tolerability of Selective Laser Trabeculoplasty vs. Pattern Laser Trabeculoplasty in Patients With Open-angle Glaucoma
Brief Title: Prospective,Randomized,Controlled Study to Assess Efficacy,Safety, and Tolerability of SLT vs. PLT in Patients With POAG
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: departure of principal investigator from the organisation
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Dr. Kaweh Mansouri, MD, University Hospital, Geneva
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1219
Record Dates: First submitted 2014-08-22; First posted 2014-09-04 (Estimated); Last update posted 2023-05-18 (Actual); Status verified 2023-05

CONDITIONS: Glaucoma and Ocular Hypertension
MeSH Terms: conditions — Glaucoma; Ocular Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pattern laser trabeculoplasty (PLT) (Experimental): Pattern laser trabeculoplasty
  Interventions: Device: Pattern laser trabeculoplasty (PLT)
- Selective laser trabeculoplasty (SLT) (Active Comparator): Selective laser trabeculoplasty (SLT)
  Interventions: Device: Selective laser trabeculoplasty (SLT)

INTERVENTIONS:
Device: Selective laser trabeculoplasty (SLT) — Selective laser trabeculoplasty
  Arms: Selective laser trabeculoplasty (SLT)
Device: Pattern laser trabeculoplasty (PLT) — Pattern laser trabeculoplasty (PLT)
  Arms: Pattern laser trabeculoplasty (PLT)

SUMMARY:
A prospective, randomized, controlled study to assess efficacy, safety, and tolerability of selective laser trabeculoplasty vs. pattern laser trabeculoplasty in patients with open-angle glaucoma.

DETAILED DESCRIPTION:
This is a prospective, randomised, controlled study. Patients will be selected for this study who require bilateral laser trabeculoplasty for IOP control. Eyes will undergo a medication wash-out 4 weeks prior to the baseline study session (S1). There will be a security visit at 2 weeks to make sure that the IOPs remain within a safe range. Following S1 both study eyes will receive laser treatment, as assigned by randomization, within a period of 2 weeks. Eyes will be randomized to receive the SLT (SLT eye) or PLT (PLT eye) treatment. Both laser procedures will be performed in one session (for 360° of the angle), if patients tolerate it. Otherwise, they will be split into two sessions (each treating 180° of the angle) to be performed within 1 week of each other. The same pre- and post-laser procedures will be applied on both eyes.

After having signed and dated the patient informed consent form, patients will undergo an initial ophthalmic examination. The CLS will be placed on both eyes for a baseline 24-hour IOP pattern recording session (S1), within 2 weeks preceding the laser treatment. Patients will remain ambulatory and will be encouraged to follow a schedule as close to his/her usual lifestyle as possible. At hour 24, patients will return to the clinic, the device will be removed and a final ophthalmic examination will be conducted. Patient diary will be collected and concomitant medication will be reported.

Following S1 both study eyes will receive either SLT or PLT laser treatment, as assigned by randomization (1:1), within a period of 2 weeks. The same pre- and post-laser procedures will be applied on both eyes.

At S2 (1 month after laser treatment) patients will be randomized to 24-hour CLS recording on either the SLT or on the PLT eye (1:1). The same ophthalmic examinations as during S1 will be conducted and patient diary collected.

At month 3 patients will be followed up with a slit lamp examination and IOP measurement. At months 6 and 12, patients will be seen for a complete ophthalmic examination including visual field exam (Octopus, Switzerland), optic nerve and retinal nerve fiber layer evaluation (Spectralis OCT, Germany). The overall study duration for the patient is limited to up to 14 months.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of open angle glaucoma (OAG) including pseudo-exfoliative and pigmentary glaucoma
* Patients requiring bilateral laser trabeculoplasty for IOP control
* Structural glaucomatous damage and/or documented glaucomatous VF damage (in the previous 12 months with mean defect (MD) > 2.5 dB
* No or stable anti-glaucomatous drug therapy since at least 3 months. Able to undergo medication washout for 4 weeks prior to baseline 24-h IOP monitoring session.
* Aged ≥18 years, of either sex
* Not more than 6 diopters spherical equivalent on the study eye
* Have given written informed consent, prior to any investigational procedures

Exclusion Criteria:

* Refractory glaucoma
* Patients having undergone ocular laser procedures (SLT, LPI) or intraocular surgery for the treatment of glaucoma.
* Corneal or conjunctival abnormality precluding contact lens adaptation
* Severe dry eye syndrome
* Patients with allergy to corneal anesthetic
* Patients with contraindications for silicone contact lens wear
* Patients not able to understand the character and individual consequences of the investigation
* Participation in other clinical research within the last 4 weeks
* Any other contra-indication listed in the CLS (SENSIMED Triggerfish) user manual

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2014-04; Primary Completion 2016-04 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
• Change in IOP from baseline to 1 month post-surgery as measured by tonometry | 1 month
  Change in IOP from baseline to 1 month post-surgery as measured by tonometry

SECONDARY OUTCOMES:
o Complete success: Reduction of at least 20% in IOP without medication | 1 month
  Complete success: Reduction of at least 20% in IOP without medication
o Qualified success: Reduction of at least 20% in IOP with IOP-lowering medication | 1 Month
  Qualified success: Reduction of at least 20% in IOP with IOP-lowering medication

OTHER OUTCOMES:
• CLS derived parameters including: o Wake-to-Sleep slopes, as measured by the linear change in IOP from before going to bed to after | 3 and 6 months
  CLS derived parameters including:

CONTACTS AND LOCATIONS:
Overall Officials: Kaweh Mansouri, Principal Investigator — Ophtalmology department - Hôpitaux Universitaires de Genève
Locations (1):
- Hôpitaux Universitaires de Genève, Ophtalmology Department, Geneva, Switzerland

REFERENCES:
- [Derived] Rolim-de-Moura CR, Paranhos A Jr, Loutfi M, Burton D, Wormald R, Evans JR. Laser trabeculoplasty for open-angle glaucoma and ocular hypertension. Cochrane Database Syst Rev. 2022 Aug 9;8(8):CD003919. doi: 10.1002/14651858.CD003919.pub3. PMID 35943114